CLINICAL TRIAL: NCT04601597
Title: Midline Catheter Tip Position and Catheter-Related Complications in Antimicrobial Therapy- A Multi-centre Randomized Controlled Trial
Brief Title: A Multicentre Pilot Study of Midline Catheter's Tip at a Different Position in Antimicrobial Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yong Fang, Director, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IVTEAM2020-01
Record Dates: First submitted 2020-09-10; First posted 2020-10-26 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Infection
Keywords: Infection nursing
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The catheter tip was placed in the subclavian vein. (Experimental): The pre-placement catheter length measured through the body surface was greater than the actual length. Therefore, 2 cm was subtracted from the pre-puncture point to the ipsilateral sternoclavicular joint to calculate the effective catheter pre-placement length.
  Interventions: Device: Shu Bei Kang (China) Midline Catheters
- The tip of the catheter was placed in the axillary vein of the chest wall. (Experimental): The pre-placement length of the catheter was measured by subtracting 3-4 cm from the distance between the puncture point and ipsilateral midclavicular line. This adjustment was intended to prevent the catheter tip from entering the subclavian vein.
  Interventions: Device: Shu Bei Kang (China) Midline Catheters
- the catheter tip was located distal to the axillary vein. (Experimental): The measurement method of catheter pre-placement length was as follows: in cases where the catheter was punctured from the basilic and brachial veins, the distance from the pre-puncture point to the intermuscular sulcus of the ipsilateral deltoid muscle and pectoralis major muscle was measured (not surpassing the intermuscular sulcus and not reaching the axilla); however, the distance from the pre-puncture point to the ipsilateral sub shoulder or axilla was measured.
  Interventions: Device: Shu Bei Kang (China) Midline Catheters

INTERVENTIONS:
Device: Shu Bei Kang (China) Midline Catheters — The procedures ① evaluation and selection of blood vessels: select the puncture vein in the middle of the patient's upper arm, ② Skin disinfection and towel laying: take the supine position, extend the upper limb to be punctured 45 ~ 90 °, disinfect the pre punctured upper limb with 75% alcohol and 5% povidone iodine. ③ Puncture vein: tie a tourniquet to fill the vein. Before puncture, use 0.2 ~ 0.4 ml of 2% lidocaine for local anesthesia. Under the guidance of ultrasound, use the puncture needle in the improved sedinger assembly for puncture. After successful puncture, insert the guide wire. ④ Delivery and confirmation of catheter position: after successful puncture, insert the dilator catheter sheath assembly, withdraw the setinger guide wire, deliver the catheter, after catheter placement, flush and seal the catheter with normal saline, and fix the catheter with sterile dressing.

SUMMARY:
The research protocol was based on assigning patients to three different catheter tip groups and then observing the relationship between the tip and catheter-related complications when infusing antimicrobial agents.

DETAILED DESCRIPTION:
A prospective case-control observation study method was adopted. The investigators of each center included patients who met the inclusion and exclusion criteria and were fully informed about the content of the study, possible benefits, and risks. After obtaining informed consent, the patients were included in the method of continuous sampling and convenient sampling. According to the method of random control, the patients were grouped. In the control group, the length of catheter insertion is measured from the pre-puncture point to the shoulder or armpit. In experimental group 1, the catheter insertion length is measured from the pre-puncture point to the midpoint of the clavicle, and in the experimental group, 2 catheter insertion length is measured from the pre-puncture point to the sternoclavicular joint. With a single-blind design, patients do not know the enrollment situation. The catheter was inserted by a full-time specialist nurse of intravenous therapy under ultrasound guidance combined with the modified Seedinger technique. The catheter was inserted according to the length of different measurement methods in different groups. After the catheter was inserted, an X-ray examination was performed to determine the catheter tip position again. Data collection and follow-up observation will be conducted by researchers who have been uniformly trained. Record the baseline data of the patients in the group before catheterization, record the insertion status during catheterization, record the patient's catheter use and catheter sealing frequency every day during catheter placement, and evaluate catheter function and complications until extubation daily.

ELIGIBILITY:
Inclusion Criteria:

Expected intravenous infusion time over 1 week In line with the indications for the use of medium-length catheters More than 18 years old Full consciousness Signed the study informed consent

Exclusion Criteria:

Source of infection at the catheter insertion site History of radiation therapy, history of thrombosis, history of trauma or vascular surgery at the site of catheterization Treatment requires input of irritating or hyperosmolar solutions Patients who need to be discharged with a catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of Phlebitis | through study completion, an average of 4 weeks
  Prolonged veins appear red, swollen, hot, and painful, with severe cord-like changes and indurations when touching. Mechanical phlebitis, infectious phlebitis, and thrombophlebitis are collected as phlebitis data
Rate of Catheter-related thrombosis | through study completion, an average of 4 weeks
  The PICC-related thrombosis in this study refers only to symptomatic thrombi, excluding asymptomatic thrombi. Catheter-related venous thrombosis was diagnosed by color Doppler ultrasound examination when the clinical manifestations were related symptoms such as swelling and pain in the upper arm of the catheterization side.
Rate of Occlusion | through study completion, an average of 4 weeks
  According to the degree, it is divided into complete occlusion and incomplete occlusion. When there is resistance or difficulty in flushing the tube, poor blood withdrawal or even no blood return can indicate that the catheter is incompletely occlusion; if it is difficult to flush the tube and draw blood, it can indicate that the catheter is completely occlusion.
Rate of Catheter-Related Infection | through study completion, an average of 4 weeks
  Including local infection of the puncture site and catheter-related blood stream infection (Catheter-Related Blood stream Infection, CRBSI). Local infection refers to redness, swelling and pain around the puncture point, or even pus; Catheter-associated bloodstream infection: refers to patients with indwelling catheters who develop bacteremia and draw blood cultures through peripheral veins for at least one positive result, accompanied by fever (> 380C), chills, or hypotension. Other clear sources of bloodstream infection.
Rate of Bleeding | through study completion, an average of 4 weeks
  Bloody fluid still leaks out of catheter puncture 48 hours after catheter insertion
Rate of Dislodgment | through study completion, an average of 4 weeks
  The catheter slipped more than 3cm above the exposed length of the first tube placement
Rate of exudation | through study completion, an average of 4 weeks
  There is a slight yellow or clear liquid leakage from the catheter puncture site

SECONDARY OUTCOMES:
Dwell time | through study completion, an average of 4 weeks
  Time from tube insertion to extubation, in days
Endometrial conditions | 24 hours before intubation and after extubation
  Ultrasound examination of the vascular intima before catheterization and within 24 hours after extubation was performed. No abnormality in the intimal smoothness was negative, and abnormalities in the intimal smoothness and hyperplasia were positive.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujiang
  - Changshu first people's Hospital, Suzhou, Jiangsu
  - Kunshan first people's Hospital, Suzhou, Jiangsu
  - Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Zhejiang Second Hospital Affiliated to Medical College of Zhejiang University, Hangzhou, Zhejiang
  - Sir Runrun Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chopra V, Kaatz S, Swaminathan L, Boldenow T, Snyder A, Burris R, Bernstein SJ, Flanders S. Variation in use and outcomes related to midline catheters: results from a multicentre pilot study. BMJ Qual Saf. 2019 Sep;28(9):714-720. doi: 10.1136/bmjqs-2018-008554. Epub 2019 Mar 18. PMID 30886119
- [Background] Xu T, Kingsley L, DiNucci S, Messer G, Jeong JH, Morgan B, Shutt K, Yassin MH. Safety and utilization of peripherally inserted central catheters versus midline catheters at a large academic medical center. Am J Infect Control. 2016 Dec 1;44(12):1458-1461. doi: 10.1016/j.ajic.2016.09.010. PMID 27908432
- [Background] Scoppettuolo G, Pittiruti M, Pitoni S, Dolcetti L, Emoli A, Mitidieri A, Migliorini I, Annetta MG. Ultrasound-guided "short" midline catheters for difficult venous access in the emergency department: a retrospective analysis. Int J Emerg Med. 2016 Dec;9(1):3. doi: 10.1186/s12245-016-0100-0. Epub 2016 Feb 4. PMID 26847572
- [Background] Paladini A, Chiaretti A, Sellasie KW, Pittiruti M, Vento G. Ultrasound-guided placement of long peripheral cannulas in children over the age of 10 years admitted to the emergency department: a pilot study. BMJ Paediatr Open. 2018 Mar 28;2(1):e000244. doi: 10.1136/bmjpo-2017-000244. eCollection 2018. PMID 29637197
- [Background] Lisova K, Hromadkova J, Pavelkova K, Zauska V, Havlin J, Charvat J. The incidence of symptomatic upper limb venous thrombosis associated with midline catheter: Prospective observation. J Vasc Access. 2018 Sep;19(5):492-495. doi: 10.1177/1129729818761276. Epub 2018 Mar 16. PMID 29546782
- [Background] Zhao Y, Geng J, Wu X, Xiong S, Wang L, Wang J, Ma H, Wei F, Wei Z. Safety of locating the tip of a medium-long catheter at the axillary front and clavicle midline: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Dec 11;99(50):e23726. doi: 10.1097/MD.0000000000023726. PMID 33327363
- [Background] Nickel B. Does the Midline Peripheral Intravenous Catheter Have a Place in Critical Care? Crit Care Nurse. 2021 Dec 1;41(6):e1-e21. doi: 10.4037/ccn2021818. PMID 34851379
- [Background] Tripathi S, Kumar S, Kaushik S. The Practice and Complications of Midline Catheters: A Systematic Review. Crit Care Med. 2021 Feb 1;49(2):e140-e150. doi: 10.1097/CCM.0000000000004764. PMID 33372744
- [Background] Bahl A, Karabon P, Chu D. Comparison of Venous Thrombosis Complications in Midlines Versus Peripherally Inserted Central Catheters: Are Midlines the Safer Option? Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029619839150. doi: 10.1177/1076029619839150. PMID 30909723
- [Background] Lu H, Yang Q, Tian B, Lyu Y, Zheng X, Xin X. A meta-analysis of the comparison of phlebitis between midline catheters and peripherally inserted central catheters in infusion therapy. Int J Nurs Pract. 2022 Apr;28(2):e12976. doi: 10.1111/ijn.12976. Epub 2021 Jun 1. PMID 34075655
- [Background] Chen W, He L, Yue L, Park M, Deng H. Spontaneous correction of misplaced peripherally inserted central catheters. Int J Cardiovasc Imaging. 2018 Jul;34(7):1005-1008. doi: 10.1007/s10554-018-1321-5. Epub 2018 Mar 12. PMID 29532310
- [Background] Passaro G, Pittiruti M, La Greca A. The fibroblastic sleeve, the neglected complication of venous access devices: A narrative review. J Vasc Access. 2021 Sep;22(5):801-813. doi: 10.1177/1129729820951035. Epub 2020 Aug 23. PMID 32830599
- [Background] Scrivens N, Sabri E, Bredeson C, McDiarmid S. Comparison of complication rates and incidences associated with different peripherally inserted central catheters (PICC) in patients with hematological malignancies: a retrospective cohort study. Leuk Lymphoma. 2020 Jan;61(1):156-164. doi: 10.1080/10428194.2019.1646908. Epub 2019 Aug 7. PMID 31387422
- [Background] Bundgaard Madsen E, Sloth E, Skov Illum B, Juhl-Olsen P. The clinical performance of midline catheters-An observational study. Acta Anaesthesiol Scand. 2020 Mar;64(3):394-399. doi: 10.1111/aas.13516. Epub 2019 Dec 22. PMID 31823342
- [Background] Chopra V, Flanders SA, Saint S, Woller SC, O'Grady NP, Safdar N, Trerotola SO, Saran R, Moureau N, Wiseman S, Pittiruti M, Akl EA, Lee AY, Courey A, Swaminathan L, LeDonne J, Becker C, Krein SL, Bernstein SJ; Michigan Appropriateness Guide for Intravenouse Catheters (MAGIC) Panel. The Michigan Appropriateness Guide for Intravenous Catheters (MAGIC): Results From a Multispecialty Panel Using the RAND/UCLA Appropriateness Method. Ann Intern Med. 2015 Sep 15;163(6 Suppl):S1-40. doi: 10.7326/M15-0744. PMID 26369828
- [Derived] Zhao L, Fan X, Zhao L, Cai Z, Jiang F, Zhao R. Midline catheter tip position and catheter-related complications in antimicrobial therapy: A multi-center randomized controlled trial. Int J Nurs Stud. 2023 May;141:104476. doi: 10.1016/j.ijnurstu.2023.104476. Epub 2023 Mar 3. PMID 36972639

DOCUMENTS (3):
  • Study Protocol (2021-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT04601597/Prot_001.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT04601597/SAP_002.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04601597/ICF_000.pdf